CLINICAL TRIAL: NCT00695591
Title: Home Sleep Testing in Neuromuscular Disease Patients
Acronym: HSTNMD
Status: Completed | Type: Observational
Sponsor: Landon Pediatric Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: LS01
Record Dates: First submitted 2008-06-03; First posted 2008-06-12 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: Neuromuscular Disease
Keywords: Home sleep testing neuromuscular disease; Neuromuscular disease patients with FEV1<50% of predicted
MeSH Terms: conditions — Neuromuscular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- 1SevereRLD,NMD: Patients with FEV1<40%
  Interventions: Other: Evaluation for Nocturnal non invasive ventilation
- 2VerySevereRLD,NMD: FEV1<30%
  Interventions: Other: Evaluation for Nocturnal non invasive ventilation
- 3NINV: FEV1<25%,on non invasive ventilation
  Interventions: Other: Evaluation for Nocturnal non invasive ventilation
- ModerateRLD,NMD: Patients with FEV1 40-50% of predicted
  Interventions: Other: Evaluation for Nocturnal non invasive ventilation

INTERVENTIONS:
Other: Evaluation for Nocturnal non invasive ventilation — Patients will be referred for evaluation for NNIV is indicated in patients with diurnal Pa,CO2 >6.0 Pa; and 2) nocturnal Sa,O2 <88% for 5 consecutive min. End tidal CO2 representing equivalent values will be referred for NNIV

SUMMARY:
Lay Summary Patients with severe neuromuscular develop hypoventilation, which leads to elevated carbon dioxide levels. Measuring only oxygen saturation levels with pulse oximetry may be inadequate. End tidal carbon dioxide levels or arterial blood gases should be measured periodically, depending on the clinical condition of the patient. A thorough review of systems will help define any problems. Patients who are hypoventilating often have elevated carbon dioxide levels at night and complain of a morning headache, restlessness or nightmares, and poor quality sleep. This may cause daytime sleepiness. Insufficient respiration with hypoxia may occur later, especially if the lung is damaged by chronic aspiration.

We propose to evaluate the use of the Nonin LifeSense monitor in home evaluation of respiration, oxygen level, heart rate, and carbon dioxide level and to develop interpretation of the results that will lead to appropriate interventions for apnea, and insufficient respiration.

Relevance to MDA Fewer than one per cent of the Muscular Dystrophy Association have pulmonologists as co-directors.Late referral of progressive restrictive lung disease leads to invasive support of respiratory failure. Early initiation of non invasive ventilation techniques requires patience on the part of the caregiver and exploration of mask interfaces and ventilation techniques. In addition, the development of new therapies, currently manifested through enhanced diagnostic accuracy, will require new signal for initiation and in the assessment of success or failure.

Aims Aim 1. To assess the utility of a small portable device (LifeSense Monitor Nonin Medical Inc. Plymouth Minnesota) with extended recording capabilty to provide accurate diagnosis of hypoventilation.

Aim 2. To provide an easily interpretable report defining sleep hypoxemia, hypercapnea, and apnea.

Aim 3. To promote early evaluation and treatment of the respiratory problems in centers that do not have pumonologists as these are essential to prognosis, whether of survival or of quality of life, in neuromuscular diseases.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of neuromuscular disease
* Must have home caregivers

Exclusion Criteria:

* No home caregiver

Ages: 8 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Study Population Description Patients from the Neuromuscular Disease Clinic at Ventura County Medical Center
  Non-Probability Sample: invitation to volunteer
  Neuromuscular Disease
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2008-07; Primary Completion 2008-09 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
1. End tidal CO2 catheter is tolerated for six hours or more | 3 months

SECONDARY OUTCOMES:
1. Interpretable data are captured for oximetry, heart rate, and end-tidal CO2 | 3 months
2. An interpretive report is generated that will guide the non-pulmonary physician in potential interventions | 6 months
2. Patients and parents are able to apply the monitors at home and a six hour data set is collected | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Chris Landon, MD, Principal Investigator — Landon Pediatric Foundation
Locations (1):
- Pediatric Diagnostic Center, Ventura, California, United States

REFERENCES:
- [Background] Shneerson JM, Simonds AK. Noninvasive ventilation for chest wall and neuromuscular disorders. Eur Respir J. 2002 Aug;20(2):480-7. doi: 10.1183/09031936.02.00404002. PMID 12212984
- [Background] Kumar SP, Sword D, Petty RK, Banham SW, Patel KR. Assessment of sleep studies in myotonic dystrophy. Chron Respir Dis. 2007;4(1):15-8. doi: 10.1177/1479972306074480. PMID 17416148
- [Background] Kirk VG, Flemons WW, Adams C, Rimmer KP, Montgomery MD. Sleep-disordered breathing in Duchenne muscular dystrophy: a preliminary study of the role of portable monitoring. Pediatr Pulmonol. 2000 Feb;29(2):135-40. doi: 10.1002/(sici)1099-0496(200002)29:23.0.co;2-#. PMID 10639204
- [Background] Birnkrant DJ, Panitch HB, Benditt JO, Boitano LJ, Carter ER, Cwik VA, Finder JD, Iannaccone ST, Jacobson LE, Kohn GL, Motoyama EK, Moxley RT, Schroth MK, Sharma GD, Sussman MD. American College of Chest Physicians consensus statement on the respiratory and related management of patients with Duchenne muscular dystrophy undergoing anesthesia or sedation. Chest. 2007 Dec;132(6):1977-86. doi: 10.1378/chest.07-0458. PMID 18079231